CLINICAL TRIAL: NCT02810691
Title: The Effect of Soluble Fiber to Reduce Post-prandial Glycemic Excursion in Adults With Cystic Fibrosis
Acronym: SOFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Canadian Cystic Fibrosis Foundation (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SOFI
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis
Keywords: Diabetes; Fiber; Supplementation; Soluble fiber; Post-prandial blood glucose; Nutrition
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soluble fiber, dose #1 (Active Comparator): Soluble fiber supplementation with dose #1 (smaller dose) of psyllium fiber.
  Interventions: Dietary Supplement: Soluble fiber supplementation
- Soluble fiber, dose #2 (Active Comparator): Soluble fiber supplementation with dose #2 (bigger dose) of psyllium fiber.
  Interventions: Dietary Supplement: Soluble fiber supplementation
- Placebo (Placebo Comparator): A 250 ml placebo solution of orange-flavored water will be drink at breakfast.
  Interventions: Dietary Supplement: Placebo (for fiber supplementation)

INTERVENTIONS:
Dietary Supplement: Soluble fiber supplementation — Two different doses of psyllium powder will be diluted in 250 ml of orange-flavored water and drink in 5 minutes before breakfast.
  Arms: Soluble fiber, dose #1; Soluble fiber, dose #2
Dietary Supplement: Placebo (for fiber supplementation) — Placebo will consist of 250 ml of orange-flavored water to be drink in 5 minutes before breakfast.
  Arms: Placebo

SUMMARY:
With improved survival, the clinical spectrum of cystic fibrosis (CF), a complex multi systemic disease, continue to evolve. A major emerging complication is CF related diabetes (CFRD) which is occurring in 40-50% of adults. Patients who develop CFRD are at increase risk of morbidity and mortality and they are also facing an increased medical burden with insulin therapy, the only recommended treatment. Accelerated decline in weight and/or pulmonary function start 2 to 4 years before CFRD onset and this period is characterized by frequent Post-Prandial Glycemic (PPG) excursions. Higher PPG excursions are associated with lower pulmonary function and it predicts future CFRD risk. To the improved nutritional status, lung function and survival of patients, the nutritional approach for patients with CF focuses on high-energy high-fat diet and a pancreatic enzyme supplementation. However, such diet also contributes to increased PPG excursions. Based on the beneficial effects of nutrition therapy to improve PPG in other forms of pre-diabetes and diabetes, extending such benefits to patients with CF is important. The investigators aim to test the feasibility and the effectiveness of a viscous fiber supplement to reduce PPG in adult patients with CF. Using a randomized crossover design, the investigators will study the impact of two doses of a viscous fiber supplement as compared to a placebo.

DETAILED DESCRIPTION:
With improved survival, the clinical spectrum of cystic fibrosis (CF), a complex multi systemic disease, continue to evolve. A major emerging complication is CF related diabetes (CFRD). CFRD is a major co-morbidity occurring in 20% of adolescents and 40-50% of adults and is mainly due to reduced insulin secretion. Patients who develop CFRD are at increase risk of morbidity and mortality and they are also facing an increased medical burden with insulin therapy, the only recommended treatment. Because accelerated decline in weight and/or pulmonary function start 2 to 4 years before CFRD onset and that this period is characterized by frequent Post-Prandial Glycemic (PPG) excursions, the role of these PPG excursions in clinical deterioration have been investigated. The investigators have shown that higher PPG excursions are associated with lower pulmonary function and others have shown that PPG excursions predicts future CFRD risk. Food overconsumption is discouraged in other forms of diabetes to avoid overweight or obesity, but also to prevent an increase in insulin demand. In contrast, nutritional approach for patients with CF focuses on high-energy high-fat diet to meet increased energy requirements. In combination with an appropriate pancreatic enzyme supplementation, this approach contributes significantly to the improved nutritional status, lung function and survival of patients. However, such diet also contributes to increased PPG excursions. Based on the beneficial effects of nutrition therapy to improve PPG in other forms of pre-diabetes and diabetes, extending such benefits to patients with CF is important. In the context of high CF treatment burden, such approach should however be simple and not inducing weight loss. The investigators aim to test the feasibility and the effectiveness of a viscous fiber supplement to reduce PPG in adult patients with CF. Using a randomized crossover design, the investigators will study the impact of two doses of a viscous fiber supplement as compared to a placebo in controlled conditions, in 22 patients, over 8 hours, at the research center with 2 standardized mixed-meals: breakfast and lunch on PPG excursions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CF
* Aged above 18 years
* CF-Impaired glucose tolerance, CF-indeterminate glucose tolerance (INDET), de-novo diabetes not requiring immediate treatment and diabetes without pharmacological treatment, based on the oral glucose tolerance test (OGTT) performed within three months of the first visit

Exclusion Criteria:

* Treated or longstanding CFRD
* Subjects taking medication or affected by conditions that could interfere with glucose metabolism in the last 6 weeks: hemoptysis, fever, IV antibiotic treatment, pregnancy and oral steroids. If a patient presents any sign of infection confirmed by a trained CF pneumologist, OGTT testing is postponed to the next medical appointment 1 months later.
* Subjects with severe gastrointestinal disease (Crohn disease, coeliac disease and recent (<1 year) history of intestinal occlusion).
* Subjects with intestinal obstruction history.
* Allergy to an ingredient in the menu.
* Corrector or potentiator prescribed within the last 6 months prior to the first visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Plasma glucose area under the curve | 3 hours

SECONDARY OUTCOMES:
Plasma insulin area under the curve | 3 hours
Incretin hormones | Each 30 minutes, up to 510 minutes, from 8h30 am to 5h00 pm
  Glucagon-like peptide, gastric inhibitory polypeptide
Side effects of the supplement | 60, 180, 300, 420 and 540 minutes after the beginning of the test
  It will be measure with gastro-intestinal symptoms visual analog scale. There will be 3 continuous scales for gastrointestinal symptoms and 5 continuous scales to evaluate the satiety. Each scale will measure 100 mm. The score is the distance measured in millimeters from the "no pain" anchor to the participant's mark.
Positive incremental area under the curve for post-prandial glucose and insulin excursions | 3 hours
Mean plasma glucose | 9 hours (over study period)
Percentage of time with plasma glucose concentration a. >8.0 mmol/L, b. >10.0 mmol/L, c. >11.0 mmol/L, and d. <4.0 mmol/L | 9 hours (over study period)
Post-meal peak plasma glucose | 3 hours after each meal
  For the breakfast and lunch

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD,PhD, Principal Investigator — IRCM
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No